CLINICAL TRIAL: NCT02156895
Title: POST MARKETING SURVEILLANCE STUDY TO OBSERVE SAFETY AND EFFICACY OF INLYTA (REGISTERED)
Brief Title: Post Marketing Surveillance Study to Observe Safety and Efficacy of Inlyta in South Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061075
Record Dates: First submitted 2014-05-06; First posted 2014-06-05 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-08

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Korean PMS of Axitinib; Metastatic RCC ; 2nd line only
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who are using Axitinib
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — based on Axitinib approval

SUMMARY:
The objective of this study is to monitor the usage of INLYTA® in real practice, including the adverse events associated with INLYTA®.

DETAILED DESCRIPTION:
Investigators can choose any patient who is within the scope of I/E criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as advanced RCC after failure of one prior systemic therapy.

Exclusion Criteria:

* Any patient who does not agree that Pfizer or companies working on behalf of Pfizer can use his/her information.
* Patients with hypersensitivity to axitinib or to any other component of INLYTA® .
* Patients under 18.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korea who has a disease for which Axitinib is indicated
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Tower, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced renal cell carcinoma (aRCC) prescribed with Inlyta (axitinib) for first time or who were already on Inlyta during study period as part of routine practice at Korean health care centers were observed. This study was to be conducted for 6 years from the approval date of 22 Aug 2012 to 21 Aug 2018. On May 2018, Ministry of Food and Drug Safety (MFDS) has granted 3 additional years for the study, for total of 9 years for the study period.
Groups:
- Inlyta: Participants with aRCC after failure of one prior systemic therapy and who were prescribed with Inlyta 1 milligram (mg) or 5 mg tablets for first time or who were already on Inlyta as part of routine practice at Korean health care centers were observed during this PMS study.
Period: Overall Study
Arm/Group | Inlyta
Started | 111
Completed | 111
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were administered Inlyta at least once and evaluated for safety related outcomes at least once.
Groups:
- Inlyta: Participants with aRCC after failure of one prior systemic therapy and who were prescribed with Inlyta 1 mg or 5 mg tablets for first time or who were already on Inlyta as part of routine practice at Korean health care centers were observed during this PMS study.
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.92 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of Advanced Renal Cell Carcinoma (aRCC) [Mean (Standard Deviation); unit: Months] — Duration of aRCC was calculated as the start date of first administration of Inlyta minus date of initial diagnosis + 1 divided by 30.4375.
  Months | 46.84 (55.21)
Number of Participants Categorized According to Cell Component of aRCC [Count of Participants; unit: Participants] — Cell component of aRCC were classified as clear cell and other.
  Participants
    Clear cell | 110
    Other | 1
Number of Participants According to Sites of Metastasis [Count of Participants; unit: Participants] — Number of participants according to the sites of metastasis including liver, lung, bone, brain, skin, lymph nodes, other and none were reported. Participants could have more than one site of metastasis.
  Participants
    Liver | 7
    Lung | 84
    Bone | 31
    Brain | 9
    Skin | 2
    Lymph nodes | 19
    Other | 23
    None | 2
Number of Participants who Underwent Primary Lesion Surgery [Count of Participants; unit: Participants] | 77
Number of Participants With Medical History [Count of Participants; unit: Participants] — Number of participants with past or present disease (medical history) were reported in this study specific characteristic.
  Participants | 101
Number of Participants With Renal Impairment [Count of Participants; unit: Participants] | 9
Number of Participants With Hepatic Impairment [Count of Participants; unit: Participants] | 4
Number of Participants With Allergic History [Count of Participants; unit: Participants] | 6
Number of Participants who Received Chemotherapy Prior to Inlyta [Count of Participants; unit: Participants] — Number of participants who received chemotherapy prior to Inlyta were reported.
  Participants | 111
Number of Participants who Received Immunotherapy Prior to Inlyta [Count of Participants; unit: Participants] — Number of participants who received immunotherapy prior to Inlyta were reported.
  Participants | 1
Number of Participants who Received Radiation Therapy Prior to Inlyta [Count of Participants; unit: Participants] — Number of participants who received radiation therapy prior to Inlyta were reported.
  Participants | 26
Number of Participants who Received Concomitant Medication [Count of Participants; unit: Participants] — Number of participants who received concomitant medication were reported.
  Participants | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs) and Serious Adverse Drug Reactions (SADRs)
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. SAE was any untoward medical occurrence that at any dose resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect. An ADR was any untoward medical occurrence attributed to Inlyta in a participant who received Inlyta. SADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to Inlyta was assessed by the physician.
Time Frame: From first dose of Inlyta or time of the participant's informed consent through the end of the observation period of the study, which included at least 28 calendar days post last dose of drug under study (observation period for the study was of 9 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Participants
  AEs | 92
  ADRs | 79
  SAEs | 14
  SADRs | 7

2. Primary Outcome: Number of Participants With Unexpected AEs, Unexpected SAEs, Unexpected ADRs and Unexpected SADRs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. SAE was any untoward medical occurrence that at any dose resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect. An ADR was any untoward medical occurrence attributed to Inlyta in a participant who received Inlyta. SADR was any SAE that is attributed to Inlyta. Relatedness to Inlyta was assessed by the physician. An unexpected AE was an AE with a difference in nature, severity, specificity, or outcome, compared to the product licensure/safety notification of the drug. Unexpected ADRs were unexpected AEs that were, in the investigator's opinion, of causal relationship to the study treatment.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Participants
  Unexpected AEs | 34
  Unexpected ADRs | 16
  Unexpected SAEs | 4
  Unexpected SADRs | 0

3. Primary Outcome: Duration of Adverse Events
Time Frame: as for outcome 1
Population: Safety analysis set included all participants who were administered Inlyta at least once and evaluated for safety related outcomes at least once. Here, "Overall Number of Participants Analyzed" signifies number of participants without missing date or month of AE onset.
Measure: Median (Full Range); unit: Days
Arm/Group | Inlyta
Number analyzed (Participants) | 49
Days | 28 [0 to 475]

4. Primary Outcome: Number of Participants With Adverse Events by Their Severity
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. Severity was graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 where, Grade 1: mild; Grade 2: moderate; Grade 3:severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. One participant may experience more than one event hence, one participant may be included in more than one category specified below.
Time Frame: as for outcome 1
Population: Safety analysis set included all participants who were administered Inlyta at least once and evaluated for safety related outcomes at least once. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Grade 1 | 68
  Grade 2 | 54
  Grade 3 | 26
  Grade 4 | 1
  Grade 5 | 2

5. Primary Outcome: Number of Participants With Adverse Events by Their Outcome
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. The outcomes of AE included recovered, recovered with sequelae, recovering, not recovered and unknown. One participant may experience more than one event hence one participant may be included in more than one category specified below.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Recovered | 61
  Recovered with sequelae | 1
  Recovering | 38
  Not recovered | 23
  Unknown | 12

6. Primary Outcome: Number of Participants With Adverse Events by Their Seriousness Criteria
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. The seriousness criteria for AEs included results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly/birth defect, other important medical event.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Results in death | 2
  Is life-threatening | 0
  Requires inpatient hospitalization or prolongation of hospitalization | 14
  Results in persistent or significant disability/incapacity | 0
  Results in congenital anomaly/birth defect | 0
  Other important medical event | 2

7. Primary Outcome: Number of Participants With Adverse Events by Their Causality to Inlyta
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship. The causality of AEs to Inlyta were assessed by physician according to the following criteria: certain, probable/likely, possible, unlikely, conditional/unclassified and unaccessible/unclassifiable. One participant may experience more than one event hence, one participant may be included in more than one category specified below.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Certain | 1
  Probable/likely | 7
  Possible | 77
  Unlikely | 35
  Conditional/unclassified | 2
  Unaccessible/unclassifiable | 1

8. Primary Outcome: Number of Participants With Adverse Events by Their Other Causality
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. If the AEs were not related to Inlyta, physicians were required to indicate the most appropriate cause of AEs from the following: disease under the study, other disease, concomitant treatment drug or non-drug and others.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Disease under the study | 4
  Other disease | 10
  Concomitant treatment drug or non-drug | 2
  Others | 26

9. Primary Outcome: Number of Participants With Adverse Events by Their Action Taken With Study Drug
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. The action taken with study drug due to AEs included discontinuation, dosage reduced, no change, unknown and not applicable. One participant may experience more than one event hence, one participant may be included in more than one category specified below.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Discontinuation | 19
  Dosage reduced | 34
  No change | 75
  Unknown | 1
  Not applicable | 8

10. Primary Outcome: Number of Participants With Adverse Events According to Demographic Characteristics
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. Number of participants with AEs classified according to the following demographic characteristics: sex: male and female; age: less than (<) 60 years, greater than or equal to (>=) 60 and < 70 years and >= 70 years; pediatric (<19 years); geriatric (>=65 years); classification: outpatient and inpatient were reported in the outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Sex: Male | 71
  Sex: Female | 21
  Age: < 60 years | 28
  Age: >= 60 years and < 70 years | 34
  Age: >= 70 years | 30
  Pediatric(< 19 years) | 0
  Geriatric(>= 65 years) | 49
  Classification: Outpatient | 86
  Classification: Inpatient | 6

11. Primary Outcome: Number of Participants With Adverse Events According to Other Baseline Characteristics
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. Number of participants with AEs classified according to the following characteristics: duration of aRCC: < 30 months, >= 30 months and < 60 months,>= 60 months; cell component of aRCC : clear cell ,other; metastasis: yes,no; site of metastasis: liver, lung, bone, brain, skin, lymph nodes, other; primary lesion surgery: done and not done; medical history: yes and no; renal impairment: yes and no; hepatic impairment: yes and no; allergic history: yes and no; prior chemotherapy: yes and no; prior immunotherapy: yes and no; prior radiation therapy: yes and no; concomitant medication: yes and no; duration of administration: < 90 days, >=90 and <180 days and >= 180 days; daily average dose: <10 and >=10 milligrams per day (mg/day).
Time Frame: as for outcome 1
Population: Safety analysis set included all participants who were administered Inlyta at least once and evaluated for safety related outcomes at least once. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. "Number Analyzed" refers to number of participants evaluable for the specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 92
Participants
  Duration of aRCC: < 30 months | 46
  Duration of aRCC: >= 30 months and < 60 months | 22
  Duration of aRCC: >= 60 months | 24
  Cell component of aRCC: Clear cell | 92
  Cell component of aRCC: Other | 0
  Metastasis: Yes | 90
  Metastasis: No | 2
  Metastasis site: Liver: number analyzed (Participants) | 90
  Metastasis site: Liver | 6
  Metastasis site: Lung: number analyzed (Participants) | 90
  Metastasis site: Lung | 67
  Metastasis site: Bone: number analyzed (Participants) | 90
  Metastasis site: Bone | 25
  Metastasis site: Brain: number analyzed (Participants) | 90
  Metastasis site: Brain | 9
  Metastasis site: Skin: number analyzed (Participants) | 90
  Metastasis site: Skin | 2
  Metastasis site: Lymph nodes: number analyzed (Participants) | 90
  Metastasis site: Lymph nodes | 19
  Metastasis site: Other: number analyzed (Participants) | 90
  Metastasis site: Other | 18
  Primary lesion surgery: Done | 65
  Primary lesion surgery: Not done | 27
  Medical history: Yes | 85
  Medical history: No | 7
  Renal impairment: Yes | 8
  Renal impairment: No | 84
  Hepatic impairment: Yes | 4
  Hepatic impairment: No | 88
  Allergic history: Yes | 5
  Allergic history: No | 87
  Prior chemotherapy: Yes | 92
  Prior chemotherapy: No | 0
  Prior immunotherapy: Yes | 0
  Prior immunotherapy: No | 92
  Prior radiation therapy: Yes: number analyzed (Participants) | 90
  Prior radiation therapy: Yes | 21
  Prior radiation therapy: No: number analyzed (Participants) | 90
  Prior radiation therapy: No | 69
  Concomitant medication: Yes | 91
  Concomitant medication: No | 1
  Duration of administration: < 90 days: number analyzed (Participants) | 91
  Duration of administration: < 90 days | 20
  Duration of administration: >= 90 days and <180 days: number analyzed (Participants) | 91
  Duration of administration: >= 90 days and <180 days | 23
  Duration of administration: >= 180 days: number analyzed (Participants) | 91
  Duration of administration: >= 180 days | 48
  Daily average dose: < 10 mg/day: number analyzed (Participants) | 91
  Daily average dose: < 10 mg/day | 32
  Daily average dose: >= 10 mg/day: number analyzed (Participants) | 91
  Daily average dose: >= 10 mg/day | 59

12. Primary Outcome: Number of Participants With Adverse Events - Multivariate Logistic Regression Analysis
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Participants | 92
Statistical Analysis 1: Comparison: Inlyta; Test type: Other; p = 0.1244, Regression, Logistic; Multiple logistic regression including total duration of treatment with Inlyta as factor; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.97 to 1.24]

13. Primary Outcome: Number of Participants With AEs and ADRs - Special Participant Population
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. An ADR was any untoward medical occurrence attributed to Inlyta in a participant who received Inlyta.
Time Frame: as for outcome 1
Population: Special participant population included geriatric participants (aged >=65 years), participants with renal or hepatic impairment who were administered Inlyta at least once. "Number Analyzed" refers to number of participants evaluable for the specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 62
Participants
  Geriatric - AEs | 49
  Geriatric - ADRs | 41
  Renal impairment - AEs: number analyzed (Participants) | 9
  Renal impairment - AEs | 8
  Renal impairment - ADRs: number analyzed (Participants) | 9
  Renal impairment - ADRs | 6
  Hepatic impairment - AEs: number analyzed (Participants) | 4
  Hepatic impairment - AEs | 4
  Hepatic impairment - ADRs: number analyzed (Participants) | 4
  Hepatic impairment - ADRs | 3

14. Primary Outcome: Number of Participants With Tumor Response Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Tumor response based on RECIST 1.1 was defined as: complete response (CR): complete disappearance of all target and non-target lesions. All lymph nodes must be non-pathological in size (<10 mm short axis); partial response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm or unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered a sign of progression; stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study and not done.
Time Frame: From first dose of Inlyta up to first documented CR, PR, PD or SD, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Participants
  Complete response (CR) | 4
  Partial response (PR) | 29
  Progressive disease (PD) | 15
  Stable disease (SD) | 51
  Not done | 12

15. Primary Outcome: Number of Participants With Objective Response
Description: Objective response (OR) was defined as the achievement of partial or complete response to therapy based on RECIST 1.1. CR: complete disappearance of all target and non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of Inlyta up to first documented CR or PR, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Participants | 33

16. Primary Outcome: Number of Participants With Objective Response According to Demographic Characteristics
Description: OR was defined as the number of participants who have a partial or complete response to therapy. CR: complete disappearance of all target and non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Number of participants with objective response categorized according to the following demographic characteristics was presented in this outcome measure: sex: male and female; age: < 60 years, >= 60 and < 70 years, >= 70 years; pediatric (<19 years); geriatric (>=65 years); classification: outpatient and inpatient.
Time Frame: From first dose of Inlyta up to first documented CR or PR, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 33
Participants
  Sex: Male | 25
  Sex: Female | 8
  Age: < 60 years | 12
  Age: >= 60 years and < 70 years | 13
  Age: >= 70 years | 8
  Pediatric(< 19 years) | 0
  Geriatric(>= 65 years) | 17
  Classification: Outpatient | 33
  Classification: Inpatient | 0

17. Primary Outcome: Number of Participants With Objective Response According to Other Baseline Characteristics
Description: OR was defined as the number of participants who have a partial or complete response to therapy. Number of participants with OR classified according to the following characteristics included duration of aRCC: < 30 months, >= 30 months and < 60 months and >= 60 months; cell component of aRCC : clear cell and other; metastasis: yes and no; site of metastasis: liver, lung, bone, brain, skin, lymph nodes and other; primary lesion surgery: done and not done; medical history: yes and no; renal impairment: yes and no; hepatic impairment: yes and no; allergic history: yes and no; prior chemotherapy: yes and no; prior immunotherapy: yes and no; prior radiation therapy: yes and no; concomitant medication: yes and no; duration of administration: < 90 days, >=90 and <180 days and >= 180 days; daily average dose: <10 and >=10 mg/day.
Time Frame: From first dose of Inlyta up to first documented CR or PR, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure. "Number Analyzed" refers to number of participants evaluable for the specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 33
Participants
  Duration of aRCC: < 30 months | 16
  Duration of aRCC: >= 30 months and < 60 months | 9
  Duration of aRCC: >= 60 months | 8
  Cell component of aRCC: Clear cell | 33
  Cell component of aRCC: Other | 0
  Metastasis: Yes | 32
  Metastasis: No | 1
  Metastasis site: Liver: number analyzed (Participants) | 32
  Metastasis site: Liver | 3
  Metastasis site: Lung: number analyzed (Participants) | 32
  Metastasis site: Lung | 26
  Metastasis site: Bone: number analyzed (Participants) | 32
  Metastasis site: Bone | 5
  Metastasis site: Brain: number analyzed (Participants) | 32
  Metastasis site: Brain | 1
  Metastasis site: Skin: number analyzed (Participants) | 32
  Metastasis site: Skin | 0
  Metastasis site: Lymph nodes: number analyzed (Participants) | 32
  Metastasis site: Lymph nodes | 8
  Metastasis site: Other: number analyzed (Participants) | 32
  Metastasis site: Other | 8
  Primary lesion surgery: Done | 27
  Primary lesion surgery: Not done | 6
  Medical history: Yes | 27
  Medical history: No | 6
  Renal impairment: Yes | 1
  Renal impairment: No | 32
  Hepatic impairment: Yes | 1
  Hepatic impairment: No | 32
  Allergic history: Yes | 1
  Allergic history: No | 32
  Prior chemotherapy: Yes | 33
  Prior chemotherapy: No | 0
  Prior immunotherapy: Yes | 0
  Prior immunotherapy: No | 33
  Prior radiation therapy: Yes: number analyzed (Participants) | 32
  Prior radiation therapy: Yes | 6
  Prior radiation therapy: No: number analyzed (Participants) | 32
  Prior radiation therapy: No | 26
  Concomitant medication: Yes | 33
  Concomitant medication: No | 0
  Duration of administration: < 90 days | 3
  Duration of administration: >= 90 days and <180 days | 11
  Duration of administration: >= 180 days | 19
  Daily average dose: < 10 mg/day | 9
  Daily average dose: >= 10 mg/day | 24

18. Primary Outcome: Number of Participants With Objective Response - Multivariate Logistic Regression Analysis
Description: OR was defined as the achievement of partial or complete response to therapy based on RECIST 1.1. CR: complete disappearance of all target and non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of Inlyta up to first documented CR or PR, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Participants | 33
Statistical Analysis 1: Comparison: Inlyta; Test type: Other; p = 0.0109, Regression, Logistic; Multiple logistic regression including total duration of treatment with Inlyta as factor; Odds Ratio (OR) = 1.11, 95% CI 2-sided [1.02 to 1.2]

19. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dose of Inlyta to first documentation of objective tumor progression, or to death due to any cause, whichever occurred first. Tumor progression was determined from tumor assessment criteria(where data meet the criteria for progressive disease [PD]), or from death report on case report forms (CRFs). PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm or unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered a sign of progression.
Time Frame: From first dose of Inlyta up to first documented tumor progression or death, whichever occurred first, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Days | 232.9 (169.23)

20. Primary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the start of Inlyta treatment to date of disease progression. If there was no progression, the case was censored as TTP at latest follow-up. Disease progression was defined as >20% increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: From first dose of Inlyta up to first documented disease progression or latest follow-up, during observation period of the study of 9 years
Population: Efficacy analysis set included all participants who had been administered Inlyta at least once.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inlyta
Number analyzed (Participants) | 111
Days | 232.9 (169.23)

ADVERSE EVENTS:
Time Frame: From first dose of Inlyta or time of the participant's informed consent through the end of the observation period of the study, which included at least 28 calendar days post last dose of drug under study (observation period for the study was of 9 years)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. Safety analysis set included all participants who had been administered Inlyta at least once and evaluated for safety related outcomes at least once.
Arm/Group | Inlyta
All-Cause Mortality (participants affected / at risk) | 2/111
Serious Adverse Events (participants affected / at risk) | 14/111
Other Adverse Events (participants affected / at risk) | 92/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inlyta (N=111)
Anaemia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 3
Death (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cellulitis (Infections and infestations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inlyta (N=111)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina unstable (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Eustachian tube patulous (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 38
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 19
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 10
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 10
Generalised oedema (General disorders) | 2
Mucosal inflammation (General disorders) | 3
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 1
Ecthyma (Infections and infestations) | 1
Endometritis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood pressure increased (Investigations) | 2
Liver function test increased (Investigations) | 1
Thyroid function test abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 15
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 4
Ejaculation failure (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02156895/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT02156895/SAP_001.pdf